CLINICAL TRIAL: NCT00001111
Title: Pharmacokinetics, Safety, Tolerance, and Activity of Nevirapine (BI-RG-587) Alone and in Combination With AZT in Mildly to Moderately Symptomatic HIV-1 Infected Children
Brief Title: A Study of Nevirapine Used Alone or in Combination With AZT in HIV-1-Infected Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Roxane Laboratories (Industry)
Purpose: Treatment
Other Study IDs: ACTG 180; 882
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Nevirapine; Zidovudine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine

SUMMARY:
Monotherapy phase: To evaluate and compare the safety, tolerance, pharmacokinetics, and preliminary activity of nevirapine administered alone in mildly to moderately symptomatic HIV-infected children ages 2 months to less than 18 years; to evaluate and compare the safety, tolerance, and pharmacokinetics of nevirapine in HIV-infected children ages 1 day to less than 2 months. Combination therapy phase: To evaluate and compare the safety, tolerance, pharmacokinetics, and preliminary activity of nevirapine administered in combination with zidovudine (AZT) in mildly to moderately symptomatic HIV-infected children ages 2 months to less than 18 years.

Compounds with reverse transcriptase inhibitory activity that are more potent and less toxic than the nucleoside analogues are needed. Nevirapine (BI-RG-587) has shown in vitro inhibitory activity against HIV-1reverse transcriptase and has shown a synergistic inhibition of HIV-1 replication when combined with zidovudine (AZT) in a plaque reduction assay.

DETAILED DESCRIPTION:
Compounds with reverse transcriptase inhibitory activity that are more potent and less toxic than the nucleoside analogues are needed. Nevirapine (BI-RG-587) has shown in vitro inhibitory activity against HIV-1 reverse transcriptase and has shown a synergistic inhibition of HIV-1 replication when combined with zidovudine (AZT) in a plaque reduction assay.

Sixty mildly to moderately symptomatic HIV-infected children (five patients in each of four age groups) will receive oral nevirapine at 1 of 3 doses for 168 days. If preliminary activity is demonstrated and toxicity is acceptable after 84 days of treatment in the three oldest age groups (ages 2 months - less than 2 years, ages 2 years - less than 13 years, and ages 13 years - less than 18 years), children ages 1 day - less than 2 months will receive one of the three doses of nevirapine. Additionally, 15 additional patients (five in each of three age groups) will receive zidovudine in combination with nevirapine. At the end of 24 weeks of combination therapy, patients discontinue zidovudine for 2 weeks while remaining on nevirapine, in order for pharmacokinetic sampling to be done. Children will be enrolled sequentially by decreasing age and increasing nevirapine dose.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* IV gammaglobulin therapy.
* Medications for PCP prophylaxis (e.g., TMP / SMX, dapsone, aerosolized and IV pentamidine).
* Fluconazole.

Patients must have:

* HIV infection. A positive Polymerase Chain Reaction (PCR) is not acceptable as the sole evidence of HIV infection. Three out of five children in each age and dose group must have a serum p24 antigen level of 70 pg/ml or greater and/or a plasma viral titer of 50 TCID/ml or greater prior to study entry.
* Ability to be followed by their original trial center for the duration of the trial.
* Consent of parent or guardian.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Lymphocytic interstitial pneumonitis if steroid-dependent or requiring supplemental oxygen or with a pretreatment paO2 < 70 mm Hg.
* Opportunistic or serious bacterial infections within 28 days prior to entry.
* Demonstrated intolerance to zidovudine prior to administration of nevirapine (in patients enrolled in the combination therapy phase of the study).
* CDC classification of P-2D (secondary infectious diseases) and/or P-2E (secondary cancers).
* Pre-existing malignancies.

Concurrent Medication:

Excluded:

* Other approved or investigational antiretroviral agents.
* All other investigational agents (except fluconazole).
* Glucocorticoids and steroid hormones.
* Dicumarol, warfarin, and other anticoagulants.
* Digitoxin.
* Valproic acid.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Isoniazid.
* Phenobarbital and other barbiturates.
* Hepatotoxic drugs.

Patients with prior participation in this trial are excluded.

Prior Medication:

Excluded:

* More than 6 weeks of prior zidovudine (AZT) therapy or more than 6 weeks of any other antiretroviral therapy.

Excluded within 7 days prior to study entry:

* AZT (in monotherapy groups only).

Excluded within 4 weeks prior to study entry:

* Other approved or investigational antiretroviral agents.
* All other investigational agents.
* Glucocorticoids and steroid hormones.
* Dicumarol, warfarin, and other anticoagulants.
* Digitoxin.
* Valproic acid.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Isoniazid.
* Phenobarbital and other barbiturates. Active alcohol or drug abuse to impair compliance with the protocol.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35
Dates: Primary Completion 1995-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Sullivan, Study Chair; K Luzuriaga, Study Chair
Locations (7):
- United States (7):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatrics, Los Angeles, California
  - Univ of Connecticut Health Ctr / Pediatrics, Farmington, Connecticut
  - Univ of Miami (Pediatric), Miami, Florida
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med Ctr / Biotech II, Worcester, Massachusetts
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey

REFERENCES:
- [Background] Luzuriaga K, Bryson Y, Krogstad P, Robinson J, Stechenberg B, Lamson M, Cort S, Sullivan JL. Combination treatment with zidovudine, didanosine, and nevirapine in infants with human immunodeficiency virus type 1 infection. N Engl J Med. 1997 May 8;336(19):1343-9. doi: 10.1056/NEJM199705083361902. PMID 9134874
- [Background] Sullivan J, Luzuriaga K. Nevirapine activity and emergence of resistant virus in pediatric trials. The ACTG 180 Study Team. Int Conf AIDS. 1993 Jun 6-11;9(1):475 (abstract no PO-B26-2042)
- [Background] Luzuriaga K, Bryson Y, McSherry G, Robinson J, Stechenberg B, Scott G, Lamson M, Cort S, Sullivan JL. Pharmacokinetics, safety, and activity of nevirapine in human immunodeficiency virus type 1-infected children. J Infect Dis. 1996 Oct;174(4):713-21. doi: 10.1093/infdis/174.4.713. PMID 8843207